CLINICAL TRIAL: NCT05622344
Title: StableEyes With Active Neurophysiological Feedback
Brief Title: StableEyes With Active Neurofeedback
Acronym: SWAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00281972; 80NSSC21M0057 (Other Grant/Funding Number: NASA)
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Vestibular Disorder; Vestibular Schwannoma; Space Motion Sickness; Motion Sickness
MeSH Terms: conditions — Vestibular Diseases; Neuroma, Acoustic; Space Motion Sickness; Motion Sickness

STUDY DESIGN:
Intervention Model Description: At each site, one group will receive the control and the second group will receive the experimental treatment (novel rehab device).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional Vestibular Physical Therapy (VPT) JHU (Active Comparator): Subjects that have had their eighth cranial nerve resected will receive traditional vestibular rehabilitation exercises at Johns Hopkins University (JHU) site.
  Interventions: Behavioral: Traditional Therapy
- SWAN VPT JHU (Experimental): Subjects that have had their eighth cranial nerve resected will receive the automated vestibular rehabilitation method
  Interventions: Device: SWAN
- SWAN Motion Sick Dayton (Experimental): Healthy control subjects that meet similar similar physical characteristics of astronauts will receive the automated vestibular rehabilitation method post motion sickness.
  Interventions: Device: SWAN
- Traditional Motion Sick Dayton (No Intervention): Typically, the suggestion for treating motion sickness once it has started is to avoid motion. Therefore, healthy control subjects that meet similar similar physical characteristics of astronauts will not receive any post motion sickness treatment.

INTERVENTIONS:
Behavioral: Traditional Therapy — Exercises that teaches subjects to move their heads while viewing still or moving targets.
  Other Names: Gaze stability exercises
  Arms: Traditional Vestibular Physical Therapy (VPT) JHU
Device: SWAN — The SWAN device uses video-oculography to monitor head motion while guiding participants to move their head in yaw, pitch, roll planes for 15 minutes. Feedback is provided regarding frequency and plane of head rotation
  Other Names: StableEyes Training Device with video-oculography
  Arms: SWAN Motion Sick Dayton; SWAN VPT JHU

SUMMARY:
The investigators have developed a self-administered rehabilitation tool that incrementally guides the user to increase head motion to mitigate motion sickness and enhance postural recovery following centrifugation or unilateral vestibular nerve deafferentation surgery.

DETAILED DESCRIPTION:
The rehabilitation device guides users to perform sinusoidal head rotations, matched to a metronome, about the yaw, pitch, and roll axes (60 sec epochs, 5 minutes per axis, 15 min total). The assessment for each axis consists of the number of completed epochs with each epoch requiring head rotations of a different amplitude. Subjects are instructed to begin with an 'easy' amplitude (i.e. small) and increase or decrease amplitude depending on the subject's perception of motion sickness - which is input from 0 (absent motion sick) to 11 (vomit) using a handheld controller. Video-oculography captures eye and head velocity as well as tracks the number of blinks and saccades, metrics that can indicate worsening nausea.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. In good general health as evidenced by medical history or diagnosed with unilateral vestibular schwannoma
4. Willing to adhere to the SWAN and/or vestibular rehabilitation regimen

Exclusion Criteria:

1. Current use of anti-nausea medication
2. Presence of cervical spine pathology that limits head motion to < 30 degrees in the horizontal or vertical plane (i.e. degenerative disc disease, rheumatoid arthritis)
3. Any orthopedic pathology that prevents walking or standing independently (i.e. recent surgery)
4. Legal blindness (20/200 or worse visual acuity)
5. Treatment using a motion sickness investigational drug or other motion sickness behavioral intervention within 30 days

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Motion sickness intensity as assessed by subjective rating | Daily for up to 4 weeks
  Subjective rating of motion sickness intensity from 0 to 10. Zero denotes absent motion sickness while 10 denote vomiting.

SECONDARY OUTCOMES:
Change in Vestibulo-Ocular Reflex (VOR) gain as measured by video-oculography | Daily for up to 4 weeks
  Ratio of eye velocity to head velocity that varies from 0 to 1.2. Normal scores are greater than 0.8.
Change in Number of blinks as measured by video-oculography | Daily for up to 4 weeks
  Increase blinking is correlated with worse motion sickness.
Change in Heart rate as measured by a monitor worn over the forearm | Daily for up to 4 weeks
  Heart rate in beats per minute will be measured using a monitor worn over the forearm.
Change in Timed Up and Go Plus | Daily for up to 4 weeks
  Time measured in seconds for a subject to stand up, step over an obstacle then walk 3M before turning around and sitting down.
Change in Foam Stance - Eyes Open | Daily for up to 4 weeks
  Time in seconds to stand on foam with eyes open. Inability to stand for less than 20 seconds is associated with 3x greater risk for falling.
Change in Foam Stance - Eyes Closed | Daily for up to 4 weeks
  Time in seconds to stand on foam with eyes closed. Inability to stand for less than 20 seconds is associated with 3x greater risk for falling.
Change in Foam Stance - Eyes Open with head motion | Daily for up to 4 weeks
  Time to seconds to stand on foam with eyes open while moving head up and down. Inability to stand for less than 20 seconds is associated with 3x greater risk for falling.
Change in Foam Stance - Eyes Closed with head motion | Daily for up to 4 weeks
  Time in seconds to stand on foam with eyes closed while moving head up and down. Inability to stand for less than 20 seconds is associated with 3x greater risk for falling.
Change in Gait speed | Daily for up to 4 weeks
  Velocity to walk 6m within a 10m marked distance, measured in meters/second. Normative data exists based on decade of age.
Change in Gait endurance | Daily for up to 4 weeks
  Distance walked in 2 minutes, measure in meters.
Change in Vertical and torsional alignment nulling test (VAN and TAN) | Daily for up to 4 weeks
  Vertical alignment nulling and torsional alignment nulling ask subjects to adjust lines to there perceived horizontal. Measured in degrees.
Change in Rod and Frame Test | Daily for up to 4 weeks
  Subjects adjust a virtual line to their perceived vertical, measured in degrees.
Change in Rod and Disk Test | Daily for up to 4 weeks
  Subjects adjust a virtual line to their perceived vertical, measured in degrees.
Change in Subjective Visual Vertical | Daily for up to 4 weeks
  Subjects adjust a virtual line to their perceived vertical, measured in degrees.
Change in Daily Activity as assessed by an activity monitor | Daily for up to 4 weeks
  Subjects wear an activity monitor on their wrist Data includes daily distance walked .

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Stewart, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Naval Medical Research Unit, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No
Currently, we have no plan to share data with other researchers

REFERENCES:
- [Background] Todd CJ, Schubert MC, Rinaudo CN, Migliaccio AA. Unidirectional Vertical Vestibuloocular Reflex Adaptation in Humans Using 1D and 2D Scenes. Otol Neurotol. 2022 Oct 1;43(9):e1039-e1044. doi: 10.1097/MAO.0000000000003684. Epub 2022 Sep 9. PMID 36075099
- See also: Patent for the rehabilitation device — https://patents.google.com/patent/US9782068B2/en
- See also: Patent for the integrated video-oculography and rehabilitation device — https://patents.google.com/patent/US10136810B2/en?q=migliaccio&inventor=schubert&oq=migliaccio+and+schubert+